CLINICAL TRIAL: NCT02603107
Title: A Phase 3, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Switching From Regimens Consisting of Boosted Atazanavir or Darunavir Plus Either Emtricitabine/Tenofovir or Abacavir/Lamivudine to GS-9883/Emtricitabine/Tenofovir Alafenamide in Virologically Suppressed HIV-1 Infected Adults
Brief Title: Study to Evaluate the Safety and Efficacy of Switching From Regimens Consisting of Boosted Atazanavir or Darunavir Plus Either Emtricitabine/Tenofovir or Abacavir/Lamivudine to Bictegravir/Emtricitabine/Tenofovir Alafenamide in Virologically Suppressed HIV-1 Infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-1878; 2015-004011-20 (EudraCT Number)
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Cobicistat; cobicistat mixture with darunavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B/F/TAF (Experimental): Randomized Phase: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) for at least 48 weeks, without regard to food.
  Extension Phase: After Week 48, participants in countries where B/F/TAF is not available will be given the option to receive B/F/TAF for up to 96 additional weeks or until the product becomes accessible to participants through an access program, or until Gilead Sciences elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: B/F/TAF
- Stay on Baseline Regimen (SBR) (Experimental): Randomized Phase: Participants remained on current antiretroviral (ARV) regimen consisting of ritonavir (RTV)-boosted or cobicistat (COBI)-boosted atazanavir (ATV) or darunavir (DRV), plus either emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) or abacavir/lamivudine (ABC/3TC) for at least 48 weeks with food.
  Extension Phase: After Week 48, participants in countries where B/F/TAF is not available will be given the option to receive B/F/TAF for up to 96 additional weeks or until the product becomes accessible to participants through an access program, or until Gilead Sciences elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: RTV; Drug: ATV; Drug: DRV; Drug: COBI; Drug: ATV/co; Drug: DRV/co; Drug: FTC/TDF; Drug: ABC/3TC; Drug: B/F/TAF

INTERVENTIONS:
Drug: RTV — 100 mg capsule coadministered orally with ATV or DRV once daily with food
  Arms: Stay on Baseline Regimen (SBR)
Drug: ATV — 300 mg capsule administered orally once daily with food
  Arms: Stay on Baseline Regimen (SBR)
Drug: DRV — 800 mg tablet administered orally once daily with food
  Arms: Stay on Baseline Regimen (SBR)
Drug: COBI — 150 mg tablet coadministered orally with ATV or DRV once daily with food
  Other Names: Tybost®; GS-9350
  Arms: Stay on Baseline Regimen (SBR)
Drug: ATV/co — 300/150 mg FDC tablet administered orally once daily with food
  Other Names: Evotaz®
  Arms: Stay on Baseline Regimen (SBR)
Drug: DRV/co — 800/150 mg FDC tablet administered orally once daily with food
  Other Names: Prezcobix®
  Arms: Stay on Baseline Regimen (SBR)
Drug: FTC/TDF — 200/300 mg FDC tablet administered orally once daily without regard to food
  Other Names: Truvada®
  Arms: Stay on Baseline Regimen (SBR)
Drug: ABC/3TC — 600/300 mg tablet administered orally once daily with or without regard to food
  Arms: Stay on Baseline Regimen (SBR)
Drug: B/F/TAF — 50/200/25 mg FDC tablet administered orally once daily without regard to food
  Other Names: Biktarvy®

SUMMARY:
The primary objective of this study is to evaluate the efficacy of switching to a fixed-dose combination (FDC) of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) versus continuing on a regimen consisting of boosted atazanavir (ATV) or darunavir (DRV) plus either emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) or abacavir/lamivudine (ABC/3TC) in HIV-1 infected adults who are virologically suppressed.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently receiving a once daily antiretroviral regimen consisting of ritonavir or cobicistat boosted ATV or DRV plus either FTC/TDF or ABC/3TC for ≥ 6 months preceding the screening visit
* Adequate renal function:

  * Estimated glomerular filtration rate ≥ 50 mL/min (≥ 0.83 mL/sec) according to the Cockcroft-Gault formula
* Life expectancy ≥ 1 year
* Currently on a stable regimen for ≥ 6 months preceding the screening visit with documented plasma HIV-1 RNA < 50 copies/mL for ≥ 6 months preceding the screening visit (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL). Prior changes in antiretroviral regimen are only allowed due to tolerability issues or for regimen simplification. Unconfirmed virologic elevations of ≥ 50 copies/mL (transient detectable viremia, or "blip") prior to screening are acceptable. (If the lower limit of detection of the local HIV-1 RNA assay is < 50 copies/mL [e.g., < 20 copies/mL], the plasma HIV-1 RNA level cannot exceed 50 copies/mL on two consecutive HIV-1 RNA tests)
* Have no documented or suspected resistance to FTC, tenofovir, ABC or 3TC, including but not limited to the reverse transcriptase resistance mutations K65R and M184V/I
* No previous use of any approved or experimental integrase strand transfer inhibitor (INSTI)

Key Exclusion Criteria:

* An opportunistic illness indicative of stage 3 HIV diagnosed within the 30 days prior to screening
* Individuals experiencing decompensated cirrhosis (eg, ascites, encephalopathy, or variceal bleeding)
* Have been treated with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids during the study (eg, corticosteroids, immunoglobulins, and other immune- or cytokine based therapies)
* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
* A history of or ongoing malignancy (including untreated carcinoma in-situ) other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma. Individuals with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of Day 1 and are not anticipated to require systemic therapy during the study
* Active, serious infections (other than HIV 1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1
* Participation in any other clinical trial, including observational studies, without prior approval from the sponsor is prohibited while participating in this trial
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the individual unsuitable for the study or unable to comply with the dosing requirements
* Any known allergies to the excipients of B/F/TAF FDC or ATV, RTV, DRV, COBI, FTC/TDF or ABC/3TC
* Females who are pregnant (as confirmed by positive serum pregnancy test)
* Females who are breastfeeding
* Acute hepatitis in the 30 days prior to study entry
* Chronic hepatitis B infection in individuals not on a TDF containing regimen, as determined by either:

  * Positive hepatitis B virus (HBV) surface antigen and negative HBV surface antibody, regardless of HBV core antibody status, at the screening visit
  * Positive HBV core antibody and negative HBV surface antibody, regardless of HBV surface antigen status, at the screening visit
* Active tuberculosis infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (90):
- United States (52):
  - Phoenix, Arizona
  - Los Angeles, California
  - Newport Beach, California
  - Oakland, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Leandro, California
  - Torrance, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Ft. Pierce, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Wilton Manors, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Macon, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Kansas City, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Buffalo, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Huntersville, North Carolina
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Longview, Texas
  - Annandale, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Australia (5):
  - Darlinghurst, New South Wales
  - Sydney, New South Wales
  - Fitzroy, Victoria
  - Melbourne, Victoria
  - Prahran, Victoria
- Belgium (2):
  - Brussels
  - Ghent
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
- Santo Domingo, Dominican Republic
- France (6):
  - Lyon
  - Nantes
  - Nice
  - Paris
  - Tourcoing
  - Tours
- Germany (8):
  - Düsseldorf, North Rhine-Westphalia
  - Berlin
  - Bonn
  - Cologne
  - Essen
  - Frankfurt
  - Hamburg
  - München
- Italy (2):
  - Milan
  - Roma
- Puerto Rico (3):
  - Ponce
  - Rio Piedras
  - San Juan
- Spain (2):
  - Madrid
  - Málaga
- United Kingdom (6):
  - Birmingham
  - Brighton
  - Edinburgh
  - Liverpool
  - London
  - Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Daar ES, DeJesus E, Ruane P, Crofoot G, Oguchi G, Creticos C, Rockstroh JK, Molina JM, Koenig E, Liu YP, Custodio J, Andreatta K, Graham H, Cheng A, Martin H, Quirk E. Efficacy and safety of switching to fixed-dose bictegravir, emtricitabine, and tenofovir alafenamide from boosted protease inhibitor-based regimens in virologically suppressed adults with HIV-1: 48 week results of a randomised, open-label, multicentre, phase 3, non-inferiority trial. Lancet HIV. 2018 Jul;5(7):e347-e356. doi: 10.1016/S2352-3018(18)30091-2. Epub 2018 Jun 18. PMID 29925490
- [Result] Andreatta K, Willkom M, Martin R, Chang S, Wei L, Liu H, Liu YP, Graham H, Quirk E, Martin H, White KL. Switching to bictegravir/emtricitabine/tenofovir alafenamide maintained HIV-1 RNA suppression in participants with archived antiretroviral resistance including M184V/I. J Antimicrob Chemother. 2019 Dec 1;74(12):3555-3564. doi: 10.1093/jac/dkz347. PMID 31430369
- [Derived] Avihingsanon A, Chetchotisakd P, Kiertiburanakul S, Ratanasuwan W, Siripassorn K, Supparatpinyo K, Martin H, Wang H, Wong T, Wang HY. Efficacy and safety of switching to bictegravir, emtricitabine, and tenofovir alafenamide in virologically suppressed Asian adults living with HIV: A pooled analysis from three international phase III randomized trials. HIV Med. 2023 Mar;24(3):290-300. doi: 10.1111/hiv.13386. Epub 2022 Aug 17. PMID 36912172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Dominican Republic, North America, Australia, and Europe. The first participant was screened on 20 November 2015. The last study visit occurred on 23 December 2019.
Pre-assignment Details: 707 participants were screened.
Groups:
- B/F/TAF: Randomized Phase: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) 50/200/25 mg fixed-dose combination (FDC) tablet orally once daily for at least 48 weeks, without regard to food.
  Extension Phase: After Week 48, participants in countries where B/F/TAF was not available were given the option to receive B/F/TAF for up to 96 additional weeks or until the product became accessible to participants through an access program, or until Gilead Sciences elected to discontinue the study in that country, whichever occurred first.
- Stay on Baseline Regimen (SBR): Randomized Phase: Participants remained on current antiretroviral (ARV) regimen consisting of ritonavir (RTV)-boosted or cobicistat (COBI)-boosted atazanavir (ATV) or darunavir (DRV), plus either emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (200/300 mg) FDC tablet or abacavir/lamivudine (ABC/3TC) (600/300 mg) FDC tablet administered orally once daily for at least 48 weeks with food.
  Extension Phase: After Week 48, participants in countries where B/F/TAF was not available were given the option to receive B/F/TAF for up to 96 additional weeks or until the product became accessible to participants through an access program, or until Gilead Sciences elected to discontinue the study in that country, whichever occurred first.
Period: Randomized Phase
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Started | 290 | 287
Completed | 275 | 266
Not Completed | 15 | 21
Not completed — Withdrew consent | 8 | 15
Not completed — Lost to Follow-up | 1 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 1
Not completed — Non-compliance with study drug | 1 | 1
Not completed — Investigator's discretion | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Optional Extension Phase
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Started | 272 (3 participants who completed the Randomized Phase did not continue in the Optional Extension Phase.) | 245 (21 participants who completed the Randomized Phase did not continue in the Optional Extension Phase.)
Completed | 263 | 232
Not Completed | 9 | 13
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrew consent | 3 | 2
Not completed — Investigator's discretion | 2 | 2
Not completed — Pregnancy | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Not treated in extension phase | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug.
Groups:
- B/F/TAF: Randomized Phase: B/F/TAF (50/200/25 mg) FDC tablet administered orally once daily for at least 48 weeks without regard to food.
  Extension Phase: After Week 48, participants in countries where B/F/TAF was not available were given the option to receive B/F/TAF for up to 96 additional weeks or until the product became accessible to participants through an access program, or until Gilead Sciences elected to discontinue the study in that country, whichever occurred first.
- Stay on Baseline Regimen (SBR): Randomized Phase: Participants remained on current ARV regimen consisting of RTV or COBI boosted ATV or DRV, plus either FTC/TDF (200/300 mg) FDC tablets or ABC/3TC (600/300 mg) FDC tablet administered orally once daily for at least 48 weeks with food.
  Extension Phase: After Week 48, participants in countries where B/F/TAF was not available were given the option to receive B/F/TAF for up to 96 additional weeks or until the product became accessible to participants through an access program, or until Gilead Sciences elected to discontinue the study in that country, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR) | Total
Number analyzed (Participants) | 290 | 287 | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10.5) | 46 (10.5) | 46 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 53 | 100
  Male | 243 | 234 | 477
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 6 | 10 | 16
  Black | 79 | 72 | 151
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  White | 188 | 190 | 378
  Other | 14 | 12 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 47 | 107
  Not Hispanic or Latino | 230 | 240 | 470
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 15 | 16 | 31
  Canada | 18 | 15 | 33
  Belgium | 2 | 3 | 5
  France | 17 | 17 | 34
  Germany | 28 | 33 | 61
  Italy | 3 | 5 | 8
  Spain | 6 | 4 | 10
  United Kingdom | 31 | 23 | 54
  United States | 166 | 164 | 330
  Dominican Republic | 4 | 7 | 11
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 285 | 277 | 562
  ≥ 50 copies/mL | 5 | 10 | 15
CD4 Cell Count [Mean (Standard Deviation); unit: cells/μL] | 669 (303.4) | 657 (285.0) | 663 (294.2)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  < 50 cells/μL | 0 | 0 | 0
  ≥ 50 to < 200 cells/μL | 4 | 8 | 12
  ≥ 200 to < 350 cells/μL | 26 | 30 | 56
  ≥ 350 to < 500 cells/μL | 62 | 60 | 122
  ≥ 500 cells/μL | 198 | 189 | 387
HIV Disease Status [Count of Participants; unit: Participants]
  Asymptomatic | 240 | 234 | 474
  Symptomatic HIV Infection | 16 | 20 | 36
  Acquired Immunodeficiency Syndrome (AIDS) | 34 | 33 | 67
Prior ARV Regimen [Count of Participants; unit: Participants]
  Boosted ATV + ABC/3TC | 21 | 23 | 44
  Boosted DRV + ABC/3TC | 24 | 21 | 45
  Boosted ATV + FTC/TDF | 105 | 110 | 215
  Boosted DRV + FTC/TDF | 140 | 133 | 273

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Determined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set: all participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- B/F/TAF: Randomized Phase: B/F/TAF (50/200/25 mg) FDC tablet administered orally once daily for at least 48 weeks without regard to food.
- Stay on Baseline Regimen (SBR): Randomized Phase: Participants remained on current ARV regimen consisting of RTV or COBI boosted ATV or DRV, plus either FTC/TDF (200/300 mg) FDC tablet or ABC/3TC (600/300 mg) FDC tablet administered orally once daily for at least 48 weeks with food.
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 290 | 287
percentage of participants | 1.7 | 1.7
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); The null hypothesis was that the percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 in the B/F/TAF group was at least 4% higher than the rate in the SBR group; the alternative hypothesis was that the percentage of participants with HIV-1 RNA ≥ 50 copies/mL in the B/F/TAF group was less than 4% higher than that in the SBR group; Test type: Non-Inferiority — A sample size of 520 participants (260 participants per treatment group) would provide at least 90% power to establish a non-inferiority margin of 4% in the Week 48 response rate (HIV-1 RNA ≥ 50 copies/mL) between the 2 treatment groups. Sample size was based on the assumptions that both treatment groups have 2% of participants with HIV-1 RNA ≥ 50 copies/mL (based on Gilead Genvoya and Stribild studies) and that the significance level of the test is at a 1-sided 0.025 level; Difference in Percentages = -0.0, 95.002% CI 2-sided [-2.5 to 2.5] — The difference in percentages and its 95.002% confidence interval (CI) were calculated based on an unconditional exact method using 2 inverted 1-sided tests
Statistical Analysis 2: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Superiority; p = 1.00, Fisher Exact

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Determined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 290 | 287
percentage of participants | 92.1 | 88.9
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Non-Inferiority — The non-inferiority of B/F/TAF would be established if the lower bound of the 2-sided 95.002% CI of the difference between the treatment groups (B/F/TAF group - SBR group) in the percentage of participants with HIV-1 RNA < 50 copies/mL is greater than -10%; Difference in Percentages = 3.2, 95.002% CI 2-sided [-1.6 to 8.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Superiority; p = 0.20, Fisher Exact

3. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 265 | 256
cells/μL | 25 (151.2) | 0 (159.4)
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Superiority; p = 0.068, ANOVA; Difference in Least Squares Means (LSM) = 25, 95% CI 2-sided [-2 to 52]

ADVERSE EVENTS:
Time Frame: From the first dose date up to last dose date (maximum: 181 weeks) plus 30 days
Description: Safety Analysis Set included participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- B/F/TAF (Randomized Phase): Randomized Phase: B/F/TAF (50/200/25 mg) FDC tablet administered orally once daily for at least 48 weeks without regard to food.
- Stay on Baseline Regimen (SBR) (Randomized Phase): Randomized Phase: Participants remained on current ARV regimen consisting of RTV or COBI boosted ATV or DRV, plus either FTC/TDF (200/300 mg) FDC tablet or ABC/3TC (600/300 mg) FDC tablet administered orally once daily for at least 48 weeks with food.
- Extension B/F/TAF From B/F/TAF; Extension B/F/TAF From SBR: After Week 48, participants in countries where B/F/TAF was not available were given the option to receive B/F/TAF for up to 96 additional weeks or until the product became accessible to participants through an access program, or until Gilead Sciences elected to discontinue the study in that country, whichever occurred first.
Arm/Group | B/F/TAF (Randomized Phase) | Stay on Baseline Regimen (SBR) (Randomized Phase) | Extension B/F/TAF From B/F/TAF | Extension B/F/TAF From SBR
All-Cause Mortality (participants affected / at risk) | 1/290 | 1/287 | 0/272 | 1/244
Serious Adverse Events (participants affected / at risk) | 17/290 | 21/287 | 20/272 | 29/244
Other Adverse Events (participants affected / at risk) | 117/290 | 126/287 | 108/272 | 113/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (Randomized Phase) (N=290) | Stay on Baseline Regimen (SBR) (Randomized Phase) (N=287) | Extension B/F/TAF From B/F/TAF (N=272) | Extension B/F/TAF From SBR (N=244)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Myxomatous mitral valve degeneration (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Optic disc disorder (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Acute hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 1
Hepatitis A (Infections and infestations) | 2 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 1 | 0
Neurosyphilis (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1
Stoma site abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Thrombotic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Physical assault (Social circumstances) | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (Randomized Phase) (N=290) | Stay on Baseline Regimen (SBR) (Randomized Phase) (N=287) | Extension B/F/TAF From B/F/TAF (N=272) | Extension B/F/TAF From SBR (N=244)
Diarrhoea (Gastrointestinal disorders) | 24 | 17 | 19 | 12
Influenza (Infections and infestations) | 7 | 12 | 10 | 15
Nasopharyngitis (Infections and infestations) | 23 | 35 | 24 | 38
Syphilis (Infections and infestations) | 9 | 11 | 14 | 14
Upper respiratory tract infection (Infections and infestations) | 23 | 24 | 24 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 16 | 12 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 19 | 15 | 13
Headache (Nervous system disorders) | 34 | 14 | 13 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 14 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Study Protocol: Original (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT02603107/Prot_004.pdf
  • Study Protocol: Amendment 1 (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT02603107/Prot_005.pdf
  • Study Protocol: Amendment 2 (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT02603107/Prot_006.pdf
  • Statistical Analysis Plan: Week 48 (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT02603107/SAP_008.pdf
  • Statistical Analysis Plan: Final (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT02603107/SAP_009.pdf